CLINICAL TRIAL: NCT05671250
Title: Novel Bioactive Smart Dressings for Diabetic Foot Ulcers: a Randomized Controlled Trial Comparing Efficacy of PRP-loaded Lyophilized Gel vs. Erythropoietin/Isosorbide Dinitrate Cryogel Scaffold vs. Standard of Care
Brief Title: Bioactive Smart Dressings for Diabetic Foot Ulcers: Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Toaa Ashraf, Assistant Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R.21.10.1492
Record Dates: First submitted 2023-01-01; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP gel and SOC-treatment (Experimental): platelet-lysate loaded lyophilized gel in addition to standard of care
  Interventions: Combination Product: PRP gel and SOC-treatment
- Trigel and SOC-treatment (Experimental): Erythropoietin/isosorbide dinitrate loaded cryogel scaffold in addition to standard of care
  Interventions: Combination Product: EPO/ISDN/UFH cryogel dressing
- standard of care alone (Active Comparator): sharp debridement, saline washing and saline dressing
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Combination Product: PRP gel and SOC-treatment — Platelet-lysate loaded sustained release thermo-gelling formulation
  Arms: PRP gel and SOC-treatment
Combination Product: EPO/ISDN/UFH cryogel dressing — Erythropoietin/Isosorbide dinitrate loaded cryogel scaffold
  Arms: Trigel and SOC-treatment
Procedure: Standard of Care — Sharp debridement, saline washing and regular saline dressing
  Arms: standard of care alone

SUMMARY:
We propose a randomized controlled study to assess the efficacy of:

1. Platelet-lysate loaded sustained release thermo-gelling formulation (Platelets-SR)
2. EPO/ISDN/UFH cryogel dressing (Trigel) As adjuncts to standard-of-care (SOC) in the treatment of chronic DFUs compared to SOC alone for patients attending the DFU outpatient clinic at the Gastroenterology Centre, Mansoura University.

DETAILED DESCRIPTION:
The tested treatments were manufactured, tested and optimized in the research laboratories of Pharmacy School, Mansoura University under ethical approval of Pharmacy School ethics committee and Medical School IRB committee.

Our primary objective is to test the hypothesis that the proposed treatments can significantly improve the wound area regression rate assessed weekly (cm2/week) for 8 weeks as compared to SOC treatment alone.

Our secondary objectives are to assess the following: the time to complete wound closure, the rate of complete wound closure and the rate of partial wound closure of ≥ 50% and ≥ 75% at end-of-treatment visit (week 8). Wound closure is confirmed when the wound remains closed at two follow up visits. The occurrence of any adverse effects either locally or systemically will be surveilled in order to assess the safety profile of the test formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age of ≥ 18
2. Type 2 Diabetes Mellitus diagnosed as per the American Diabetic Association at the time of recruitment
3. Patients with glycated haemoglobin (HbA1C) ≤ 9% within 4 weeks prior to randomization
4. Patients with ulcer that meets the following criteria

   1. Ulcers classified as Grade 1, stage A (1A) ulcers using University of Texas (UT) classification system (ulcers are superficial not involving tendon, capsule or tendon and are non-infected and non-ischemic)
   2. Ulcer duration of 4 weeks or longer and hard to heal despite standard of care treatment (chronic ulcers)
   3. Ulcer has undergone recent debridement (2 weeks prior to screening)
   4. Post-debridement ulcer is free of necrotic debris, foreign bodies, sinus tracts, tunnelling, and undermining and is comprised of healthy vascularized tissue
   5. Wound area at start of treatment between 2 sq.cm. and 10 sq.cm.
   6. No surgical revascularization of the limb with the DFU was done in the previous two months.
5. Limb criteria: At least moderate blood perfusion into the affected limb as defined by Ankle Brachial Index (ABI) of 0.9 - 1.3.
6. Patients who agree to conform to the off-loading requirements
7. Provide written informed consent prior to admission into the study

Exclusion Criteria:

1. Type 1 Diabetes Mellitus
2. Patients who have undergone, in the 2-week period prior to enrolment, treatment for DFU with any advanced treatment modality other than standard of care, such as growth factors, skin substitutes or other biological treatments
3. Have a glycosylated haemoglobin (HbA1c) > 9.0%
4. Have a body mass index (BMI) > 40 Kg/m2
5. Have a clinically significant cardiac, gastrointestinal, endocrine, neurological, liver, or kidney disease
6. Anaemia (Haemoglobin < 9 g/dL) or white Blood Cells count > 11,000/μL or platelets count < 100,000/μL or > 400,000/μL or liver function tests > 3 times upper normal lab values or Creatinine > 3 mg/dL; any indication of malnourishment (Albumin < 3 g/dL); INR > 2 or any other clinically significant blood and urinalysis tests per the physician's discretion
7. Patients with haemochromatosis or unstable hypertension
8. Have any clinically significant chronic or acute illness during the 4 weeks prior to admission into the study, except type 2 diabetes or during screening period
9. Patients with wounds caused by basal cell carcinoma or due to basal cell carcinoma excision
10. Females who are pregnant, lactating, of child-bearing potential, or post-menopausal for less than 2 years, not using a medically approved method of contraception, or females who test positive on a blood-based pregnancy test.
11. Patients with a history of allergy to one of tested components
12. Patients on glyceryl trinitrate or Sildenafil treatment
13. Patients with a history of any clinical or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of the investigational agent or may confound the interpretation of study results or might render the patient at high risk for treatment complications
14. Patients with active Charcot or other structural deformity that would prevent adequate off-loading of the study foot.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Wound area regression rate | 8 weeks
  wound area regression rate assessed weekly (cm2/week)

SECONDARY OUTCOMES:
rate of complete wound closure | 8 weeks
  rate of complete wound closure (100% closure)
rate of partial wound closure of ≥ 75% | 8 weeks
  rate of partial wound closure of ≥ 75%
rate of partial wound closure of ≥ 50% | 8 weeks
  rate of partial wound closure of ≥ 50%

OTHER OUTCOMES:
Adverse effects | 8 weeks
  rate of adverse effects related to any of the interventions used

CONTACTS AND LOCATIONS:
Overall Officials: Toaa Ashraf, Study Director — Mansoura University; Amira Motawea, Study Director — Mansoura University; Marwa S. El-Dahhan, Study Director — Mansoura University; Fady Azmy, Study Director — Mansoura University; Galal M. Abdelghani, Principal Investigator — Mansoura University
Locations (1):
- Toaa Ashraf, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No